CLINICAL TRIAL: NCT06309069
Title: Calcified Cerebral Embolism: a Descriptive Study in a Large Single Center Cohort
Acronym: CCE Cohorte
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2024/TP-01; IRB 24.01.01 (Other: IRB)
Record Dates: First submitted 2024-02-26; First posted 2024-03-13 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Calcified Cerebral Embolism
Keywords: calcified cerebral embolism; cerebral infarction; radiological characteristics
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CCE: CCE patients identified between 2015 and 2023
  Interventions: Other: None, purely observational study

INTERVENTIONS:
Other: None, purely observational study — None, purely observational study

SUMMARY:
Calcified cerebral embolism (CCE) is a relatively rare but underdiagnosed cause of infarction. CCE diagnosis is made by CT. Radiological characteristics of CCE have been reported in small case series. The aim of this study was to describe clinical and radiological characteristics of CCE in a large number of patients, and to compare patients with different radiological CCE characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CEE treated with intravenous thrombolysis (IVT) between 2015 and 2020 managed at the CHU de Nîmes or Patients with TIA/stroke with ECC identified on CT between 12/2019 and 04/2023 managed at CHU de Nîmes

Exclusion Criteria:

* Patient's refusal to use his/her data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with CEE treated with intravenous thrombolysis (IVT) between 2015 and 2020, and patients with AIT/stroke with a CCE identified on CT between deceber 2019 and april 2023.
Sampling Method: Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Calcified aortic brachiocephalic | baseline
  looking for calcified aortic brachiocephalic (presence or absence)
cardiovascular risk | baseline
  Study of cardiovascular risk factors (presence or absence)
history of stroke | baseline
  Presence of a history of stroke (y/n)
Population | baseline
  demographic characteristics age (years)
Population | baseline
  demographic characteristics sexe (M/F)
history of surgical/endovascular cardiovascular intervention | baseline
  surgical/endovascular cardiovascular intervention (y/n)
NIHSS | baseline
  NIHSS score (Score between 1 and 4: minor stroke, Score between 5 and 15: moderate, stroke, Score between 15 and 20: severe stroke) Score > 20: severe stroke
calcified aortic arch | baseline
  looking for calcified aortic arch (presence/absence)
calcified carotid | baseline
  looking for calcified carotid (presence/absence)
atherosclerotic plaques | baseline
  looking for atherosclerotic plaques (presence/absence)
calcified aortic valves | baseline
  looking for calcified aortic valves (presence/absence)
calcified mitral valves | baseline
  looking for calcified mitral valves (presence/absence)
CCE diameter | baseline
  CCE diameter measurement (mm)
density | baseline
  CCE density (uh)
involved cerebral artery | baseline
  description of involved cerebral artery

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Result] Serghine Y, Laurent-Chabalier S, Thouvenot E, Parvu T, Renard D. Clinical and radiological characteristics of calcified cerebral embolism: a large case series including 242 calcified cerebral embolism. Acta Neurol Belg. 2025 Apr;125(2):463-468. doi: 10.1007/s13760-025-02719-w. Epub 2025 Jan 15. PMID 39813005